CLINICAL TRIAL: NCT00932139
Title: Neural Mechanism of the Effect of Acupuncture on Hypertension
Brief Title: Effect of Electro-Acupuncture on Blood Pressure
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Irvine (Other)
Responsible Party: Principal Investigator, Shaista Malik, Professor, University of California, Irvine
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 1999-2222
Record Dates: First submitted 2009-07-01; First posted 2009-07-03 (Estimated); Last update posted 2025-04-15 (Actual); Status verified 2025-04

CONDITIONS: Hypertension
Keywords: Hypertension; blood pressure; mild to moderate hypertension
MeSH Terms: conditions — Hypertension | interventions — Blood Pressure

STUDY DESIGN:
Intervention Model Description: Two different formulated sets of acupoints will be used as EA intervention in the treatment of hypertension.
Who Masked: Care Provider, Investigator, Outcomes Assessor
Masking Description: The care provider or acupuncturist does not know the outcome of the treatment. The investigator does not know the participants and the outcome of the study. The outcome assessor does not know the participants.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Electro-acupuncture control (Experimental): Blood pressure will be recorded before and after each EA treatment for 8 weeks. The course is a once a week 8-week treatment.
  Intervention is the Electro-acupuncture control treatment.
  Interventions: Procedure: Electro-acupuncture control; Procedure: Electro-acupuncture test
- Electro-acupuncture test (Experimental): Blood pressure will be recorded before and after each EA treatment for 8 weeks. The course is a once a week 8-week treatment.
  Intervention is the active Electro-acupuncture treatment.
  Interventions: Procedure: Electro-acupuncture control; Procedure: Electro-acupuncture test

INTERVENTIONS:
Procedure: Electro-acupuncture control — First visit, blood pressure monitoring for 60 minutes at rest, then monitoring for subsequent 24 hours to measure BP and heart rate. At next 6-8 visits, Electro-acupuncture (EA) treatment for 30 minutes will be administered. BP and heart rate measurements will be taken 30 minutes before and after EA.
  Other Names: Blood pressure; Hypertension
Procedure: Electro-acupuncture test — First visit, blood pressure monitoring for 60 minutes at rest, then monitoring for subsequent 24 hours to measure BP and heart rate. At next 6-8 visits, Electro-acupuncture (EA) treatment for 30 minutes will be administered. BP and heart rate measurements will be taken 30 minutes before and after EA. At end of 8-week treatment, 24 hours blood pressure and heart rate will be measured.
  Other Names: Blood pressure; Hypertension

SUMMARY:
Based on previous published research in animals and human, the investigators hypothesize that electroacupuncture (EA) will have a positive effect on hypertension.

DETAILED DESCRIPTION:
The purpose of this study is to prove: (1) hypertensive response at rest and provoked by stress are decreased by EA; (2) The mechanisms of EA that reduces elevated blood pressure. EA inhibits the sympathetic nervous system, decreases blood pressure and reduces the oxygen demand. Our prior data in animals shows that improvements in cardiovascular function during myocardial ischemia, reflex hypertension and sustained hypertension are mediated by an EA-induced sensory neural reflex originating in somatic nerves to reduce sympathetic nerve activity. The specific aims of the present study will allow us to better understand and modulate the sympathetic nervous discharge activity that can cause hypertension during normal activity and stress in humans. The potential clinical application is the therapeutic value of EA in patients with hypertension.

Furthermore, the study will also investigate gender differences in the blood pressure lowering effect of EA. In particular in middle-aged hypertensive women and men.

ELIGIBILITY:
Inclusion Criteria:

* Patients with mild coronary disease, and no significant ECG change reflecting ischemia at rest.
* Patients with high blood pressure with or without antihypertensive medication.

Exclusion Criteria:

* Pregnant or nursing women
* Individuals with severe coronary disease (continuous angina)
* Conduction abnormalities on ECG consistent with left bundle branch block
* Cardiac arrhythmias associated with low blood pressure (90 mmHg)
* Peripheral vascular disease
* Orthopedic disease
* Diabetic or psychological illness that could interfere with safe performance of exercise of psychophysiological stress testing
* Those with known sensitivity to topical preparations or strong reactions to medical dressings and skin tapes

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2003-02; Primary Completion 2027-09 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
blood pressure | 8 weeks
  evaluation of systolic and diastolic blood pressures changes

SECONDARY OUTCOMES:
Heart rate | 8 weeks
  evaluation of heart rate change
plasma catecholamine | 8 weeks
  evaluation of plasma catecholamine (ng/ml) change
plasma renin | 8 weeks
  evaluation of plasma renin (ng/ml.hr) change

CONTACTS AND LOCATIONS:
Overall Officials: Shaista Malik, MD, PhD, MPH, Principal Investigator — University of California, Irvine; Liang-Wu Fu, MD, PhD, Principal Investigator — University of California, Irvine; LiFang Xie, PhD, LAc, Principal Investigator — University of California, Irvine
Locations (2):
- United States (2):
  - Susan Samueli Integrative Health Institute, Irvine, California
  - UCIMedical Center, Orange, California

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Li P, Tjen-A-Looi SC, Cheng L, Liu D, Painovich J, Vinjamury S, Longhurst JC. Long-Lasting Reduction of Blood Pressure by Electroacupuncture in Patients with Hypertension: Randomized Controlled Trial. Med Acupunct. 2015 Aug 1;27(4):253-266. doi: 10.1089/acu.2015.1106. PMID 26392838